CLINICAL TRIAL: NCT00240994
Title: A Phase II Exploratory Study to Determine the Safety and Study the Immunomodulatory Functions of Induction Therapy With Campath, Combined With Chronic Immunosuppression With Mycophenolate Mofetil and Sirolimus
Brief Title: Safety in Immunomodulatory Functions of Alemtuzumab (Campath) in Pediatric Kidney Transplantation Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Cooperative Clinical Trials in Pediatric Transplantation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAIT PC01
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Failure, Chronic; Kidney Transplantation; Immunosuppression
Keywords: End stage renal disease; Kidney transplantation; Renal transplantation; Kidney failure; Pediatric renal transplant recipients; Alemtuzumab; Campath; Mycophenolate mofetil; MMF; CellCept; Tacrolimus; Prograf; Sirolimus; Rapamycin
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Alemtuzumab; Tacrolimus; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Campath) (Experimental): In this open-label, single-arm trial , participants will be administered a 0.3 mg/kg dose of alemtuzumab (Campath) intravenously one day prior to kidney transplantation and one day post kidney transplantation. Participants will then receive a maintenance immunosuppressive regimen of tacrolimus and mycophenolate mofetil (MMF) for 8 to 12 weeks, followed by sirolimus and MMF until 24 months post transplantation.
  Interventions: Drug: Alemtuzumab; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Sirolimus

INTERVENTIONS:
Drug: Alemtuzumab — Administered intravenously over a period of 2-3 hours. Two doses total, the first will be one day before transplant and the second will be on the day following transplantation. Pre-medication with methylprednisolone, acetaminophen, and Benadryl will be administered before each dose.
  Other Names: Campath; Campath- 1H
Drug: Tacrolimus — Administered orally at a dose of 0.05-0.1 mg/kg twice daily, beginning 1-3 days following transplantation and continuing until weeks 8-12. Tacrolimus will be discontinued and a treatment regimen with sirolimus will be initiated between weeks 8-12 but some overlap with these medications is possible.
  Other Names: Prograf
Drug: Mycophenolate mofetil — Per recommendation
  Other Names: CellCept
Drug: Sirolimus — Administered by either liquid or tablet every 12 hours from month 6 until month 24. Dosage will vary throughout the treatment course.
  Other Names: Rapamycin

SUMMARY:
The purpose of this study is to evaluate the safety of alemtuzumab after kidney transplantation as part of a multitherapy regimen to prevent kidney graft loss and death and to avoid steroids and chronic use of calcineurin inhibitors in pediatric renal transplant recipients 1 to 20 years of age.

DETAILED DESCRIPTION:
Kidney transplantation is widely considered to be the treatment of choice for children with End Stage Renal Disease (ESRD). Improvements in surgical techniques, donor selection, and immunosuppression practices, as well as the enhanced experience of specialized pediatric transplant teams, have all led to marked improvements in patient and kidney graft survival in infants and young children ages 1 to 10. However, young children now have more infections following transplant previously. Also, improved graft survival is not observed in pediatric renal transplant recipients 11 to 17 years of age. Some studies do indicate that the poor long term outcome of patient and kidney survival observed in this age group may be caused by noncompliance with immunosuppressive medications. Therefore, protocols that minimize the use of immunosuppressive medications while retaining kidney function are necessary for improving graft and patient survival in children. This study will evaluate the safety of a regimen containing alemtuzumab after kidney transplantation, followed by steroid avoidance and calcineurin inhibitor withdrawal in pediatric renal transplant recipients 1 to 20 years of age.

The accrual period is scheduled for 18 months. The study follow-up period will last 24 months. All participants enrolled will undergo this treatment schedule: 1.) All participants will receive intravenous alemtuzumab one day before transplantation and 1 day after transplantation. 2.) Mycophenolate mofetil (MMF) will be administered orally no later than 2 days after transplantation. 3.) Participants will begin to take oral tacrolimus twice a day 1 to 3 days after transplantation until Weeks 8 through 12 when 4.) Sirolimus will be initiated. 5.) Sirolimus and MMF will be taken orally until Month 24.

Blood collection will occur at baseline, 1 day before transplant, at Days 1 and 3, at Weeks 2, 4, 6, 8, 10, and at Months 3 through 24. Scheduled kidney (renal) biopsies will be performed at transplant, during Weeks 8 through 12, immediately before conversion to sirolimus, and at Months 6 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 1 to 20 (prior to 21st birthday)
* End Stage Renal Disease
* Necessity of kidney transplant
* First kidney transplant received from a living donor
* A living kidney donor identified
* No known contraindications to therapy with alemtuzumab
* Negative pregnancy test before study entry
* Willing to use approved methods of contraception for the duration of the study, 6 weeks after discontinuation of MMF, and 12 weeks after discontinuation of sirolimus
* Informed consent from participant, parent, or guardian
* Current vaccinations, including varicella-zoster (VZV) vaccine, before study enrollment

Exclusion Criteria:

* Recipient of a deceased donor kidney transplant
* Multiorgan transplant
* History of prior organ transplantation
* Participant sensitized to greater than 0% Panel Reactive Antibody (PRA) within 4 weeks before study enrollment. (If participant receives a blood transfusion status post PRA test, then the PRA must be repeated within 1 week of transplantation)
* Participants with human leukocyte antigen (HLA) identical living related donors
* History of primary focal segmented glomerulosclerosis
* History of other disorders requiring continuous maintenance steroids or calcineurin inhibitors
* Active systemic infection at time of transplant
* History of malignancy
* Infected with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Contraindication to receive tacrolimus, sirolimus, MMF, or monoclonal antibody therapy
* Use of investigational drugs within 4 weeks before study enrollment
* Recipient of any licensed or investigational live attenuated vaccine(s) within 2 months before study enrollment
* Family history of high cholesterol

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2005-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Harmon, MD, Study Chair — Boston Children's Hospital
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital, Boston, Boston, Massachusetts
  - Children's Hospital, Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital and Regional Medical Center, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Wolff G, Strecker K, Vester U, Latta K, Ehrich JH. Non-compliance following renal transplantation in children and adolescents. Pediatr Nephrol. 1998 Nov;12(9):703-8. doi: 10.1007/s004670050531. PMID 9874312
- [Background] Ciancio G, Burke GW, Gaynor JJ, Mattiazzi A, Roohipour R, Carreno MR, Roth D, Ruiz P, Kupin W, Rosen A, Esquenazi V, Tzakis AG, Miller J. The use of Campath-1H as induction therapy in renal transplantation: preliminary results. Transplantation. 2004 Aug 15;78(3):426-33. doi: 10.1097/01.tp.0000128625.29654.eb. PMID 15316372
- [Background] Rao V, Pirsch JD, Becker BN, Knechtle SJ. Sirolimus monotherapy following Campath-1H induction. Transplant Proc. 2003 May;35(3 Suppl):128S-130S. doi: 10.1016/s0041-1345(03)00227-6. PMID 12742484
- [Background] Kreis H, Cisterne JM, Land W, Wramner L, Squifflet JP, Abramowicz D, Campistol JM, Morales JM, Grinyo JM, Mourad G, Berthoux FC, Brattstrom C, Lebranchu Y, Vialtel P. Sirolimus in association with mycophenolate mofetil induction for the prevention of acute graft rejection in renal allograft recipients. Transplantation. 2000 Apr 15;69(7):1252-60. doi: 10.1097/00007890-200004150-00009. PMID 10798738
- [Background] Watson CJ, Bradley JA, Friend PJ, Firth J, Taylor CJ, Bradley JR, Smith KG, Thiru S, Jamieson NV, Hale G, Waldmann H, Calne R. Alemtuzumab (CAMPATH 1H) induction therapy in cadaveric kidney transplantation--efficacy and safety at five years. Am J Transplant. 2005 Jun;5(6):1347-53. doi: 10.1111/j.1600-6143.2005.00822.x. PMID 15888040
- [Result] De Serres SA, Mfarrej BG, Magee CN, Benitez F, Ashoor I, Sayegh MH, Harmon WE, Najafian N. Immune profile of pediatric renal transplant recipients following alemtuzumab induction. J Am Soc Nephrol. 2012 Jan;23(1):174-82. doi: 10.1681/ASN.2011040360. Epub 2011 Nov 3. PMID 22052056
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY134 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY134 — ImmPort study identifier is SDY134
- Available data/document: Study Protocol: SDY134 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY134 — ImmPort study identifier is SDY134
- Available data/document: Study summary, - schedule of events, -download packages et al.: SDY134 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY134 — ImmPort study identifier is SDY134

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four centers in the United States recruited 35 subjects between January 2005 and October 2007 who were less than 21 years of age and first time living-donor kidney allograft recipients.
Pre-assignment Details: At a screening visit, participants underwent procedures to establish inclusion/exclusion criteria and then sign the informed consent form.
Groups:
- Alemtuzumab (Campath): In this open-label, single-arm trial, participants were administered a 0.3 mg/kg dose of alemtuzumab intravenously one day prior to kidney transplantation and one day post kidney transplantation. Participants were then administered a maintenance immunosuppressive regimen of tacrolimus and mycophenolate mofetil (MMF) for 8 to 12 weeks, followed by sirolimus and MMF until 24 months post transplantation.
Period: Overall Study
Arm/Group | Alemtuzumab (Campath)
Started | 35
Completed | 32
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Graft failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab (Campath)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years]
  Final status: Completed (N=22) | 13.1 (5.0)
  Final status: Discontinued Therapy (N=10) | 9.8 (6.2)
  Final status: Discontinued Study (N=3) | 17.7 (2.4)
  All Participants (N=35) | 12.6 (5.5)
Gender [Count of Participants; unit: Participants]
  Female | 20
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants With Graft Loss or Death Within 12 Months Post Kidney Transplantation
Description: Graft loss is defined as the need for dialysis for more than 30 days duration, allograft nephrectomy, or the decision to withdraw immunosuppression due to graft failure.
Time Frame: Up to one year post kidney transplantation procedure
Population: Intent-to-treat
Measure: Number; unit: Proportion of participants
Arm/Group | Alemtuzumab (Campath)
Number analyzed (Participants) | 35
Proportion of participants | 0.057
Statistical Analysis 1: Comparison: Alemtuzumab (Campath); The proportion of participants with graft loss or death within 12 months post kidney transplantation is descriptively summarized with a 95% confidence interval using an exact binomial method; Test type: Superiority or Other; 95% Confidence Interval; 95% CI using an exact binomial method; Proportion with graft loss or death = .057, 95% CI 2-sided [0.007 to 0.192]

ADVERSE EVENTS:
Time Frame: From beginning of study to end of study
Description: This study graded the severity of adverse events experienced by the study participants according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Groups:
- Alemtuzumab (Campath): In this open-label, single-arm trial , participants were administered a 0.3 mg/kg dose of alemtuzumab intravenously one day prior to kidney transplantation and one day post kidney transplantation. Participants were then administered a maintenance immunosuppressive regimen of tacrolimus and mycophenolate mofetil (MMF) for 8 to 12 weeks, followed by sirolimus and MMF until 24 months post transplantation.
Arm/Group | Alemtuzumab (Campath)
Serious Adverse Events (participants affected / at risk) | 25/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (Campath) (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Graft loss (Immune system disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 2 (2)
Transplant rejection (Immune system disorders) | 3 (4)
Adenovirus infection (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Central line infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (4)
Herpes simplex (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (3)
Rhinovirus infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 4 (6)
Blood culture positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Epiphyseal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Glomerulonephritis focal (Renal and urinary disorders) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Gastrostomy closure (Surgical and medical procedures) | 1 (1)
Suture removal (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab (Campath) (N=35)
Anaemia (Blood and lymphatic system disorders) | 20 (35)
Leukopenia (Blood and lymphatic system disorders) | 23 (70)
Lymphopenia (Blood and lymphatic system disorders) | 4 (6)
Neutropenia (Blood and lymphatic system disorders) | 14 (26)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anal ulcer (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 12 (15)
Mouth ulceration (Gastrointestinal disorders) | 5 (11)
Nausea (Gastrointestinal disorders) | 3 (4)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 3 (4)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 7 (9)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Transplant rejection (Immune system disorders) | 2 (3)
Bronchitis (Infections and infestations) | 2 (2)
Bronchitis acute (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Chronic sinusitis (Infections and infestations) | 2 (2)
Cystitis klebsiella (Infections and infestations) | 4 (8)
Ear infection (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Impetigo (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (8)
Urinary tract infection enterococcal (Infections and infestations) | 3 (6)
Viraemia (Infections and infestations) | 3 (4)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Post procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Blood cholesterol increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 5 (7)
Blood parathyroid hormone increased (Investigations) | 3 (3)
Blood pressure increased (Investigations) | 2 (2)
Epstein-Barr virus antibody positive (Investigations) | 3 (3)
Haematocrit decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 5 (9)
Neutrophil count decreased (Investigations) | 2 (3)
Transferrin saturation decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Food intolerance (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 (8)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 3 (3)
Hypercalciuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 5 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No